CLINICAL TRIAL: NCT02271204
Title: Post Authorization Safety Study of iv Ibandronate (Bonviva) in Postmenopausal Osteoporosis, Observational, Non-interventional Open Label Trial
Brief Title: Observational Study of iv Ibandronate in Women With Postmenopausal Osteoporosis
Status: Completed | Type: Observational
Sponsor: Clinic of Endocrinology and Metabolic Disorders, Macedonia (Other)
Collaborators: Clinic for Orthopedic Surgery, Skopje (Unknown); General Hospital, Kumanovo (Unknown); General Hospital, Struga (Unknown); Medical Faculty, Institute for Epidemiology and Biostatistics, Skopje (Unknown)
Responsible Party: Sponsor
Other Study IDs: ML21741
Record Dates: First submitted 2014-10-07; First posted 2014-10-22 (Estimated); Last update posted 2014-10-22 (Estimated); Status verified 2014-10

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Ibandronic Acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Ibandronic acid — As prescribed by physician
  Other Names: Bonviva

SUMMARY:
This observational study assess the safety of intravenous Ibandronate (Bonviva) intermittent administration in patients with postmenopausal osteoporosis and the efficacy of IV Ibandronate (Bonviva treatment through relative lumbar spine and hip bone mineral densitometry form baseline at year 1)

ELIGIBILITY:
Inclusion Criteria:

* Patients had post menopausal osteoporosis
* Patients had no contraindication for bisphosphonates
* Patients had been naive for ibandronate therapy
* Patients who have signed informed consent and are willing to share their data for data analysis

Exclusion Criteria:

* Is not Ibandronate naïve
* Hypersensitivity to any component of the bisphosphonates Ibandronate;
* Administration of any investigational drug within 30 days preceding the first dose of the study drug.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with postmenopausal osteoporosis in everyday routine practice from selected centers in R. Macedonia
Sampling Method: Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2009-03; Primary Completion 2013-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events and Serious Adverse Events as a Measure of Safety and Tolerability of intravenous Ibandronate intermittent administration in patients with postmenopausal osteoporosis | end of observation 12 months